CLINICAL TRIAL: NCT05042895
Title: Hysteroscopic Findings in Ovarian Polycystic and Unexplained Infertile Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCO
Record Dates: First submitted 2021-05-23; First posted 2021-09-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A cross-sectional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCO women (Active Comparator): Group A will consist of 100 PCO infertile women
  Interventions: Procedure: Group A
- unexplained infertile cases (Active Comparator): group B will consist of 50-unexplained infertility.
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group A — Office diagnostic hysteroscopy for assessment of the following:
  * cervical canal: arborvitae, mucous, any abnormal pathology like a polyp.
  * Endometrium cavity: vascularity, thickness, color, gland openings, any abnormal pathology.
  * Darwishhysterscopic triad: shape, caliber, depth, abnormal pathology, flow patency, bubble flow patency, and peristalsis.
  Endometrial sample by a Novak's curette Histopathologic assessment: will be sent for the routine out-patient Pathology lab to comment on the endometrial pattern and abnormalities.
  Physical and laboratory examinations follicle-stimulating hormone [FSH], LH, thyroid-stimulating hormone [TSH], prolactin, and pre ovulatory LH LH levels of the patients will be measured on day 3 of the menstrual cycle.
  Other Names: Polycystic infertile women
  Arms: PCO women
Procedure: Group B — Office diagnostic hysteroscopy for assessment of the following:
  * cervical canal: arborvitae, mucous, any abnormal pathology like a polyp.
  * Endometrium cavity: vascularity, thickness, color, gland openings, any abnormal pathology.
  * Darwishhysterscopic triad: shape, caliber, depth, abnormal pathology, flow patency, bubble flow patency, and peristalsis.
  Endometrial sample by a Novak's curette Histopathologic assessment: will be sent for the routine out-patient Pathology lab to comment on the endometrial pattern and abnormalities.
  Physical and laboratory examinations follicle-stimulating hormone [FSH], LH, thyroid-stimulating hormone [TSH], prolactin, and pre ovulatory LH LH levels of the patients will be measured on day 3 of the menstrual cycle.
  Other Names: Unexplained infertility
  Arms: unexplained infertile cases

SUMMARY:
In many PCO infertile patients, abnormal endometrial echogenicity and thickness are documented by TVS and proved by endometrial biopsy in some cases. Should patients with normal appearance of the endometrium (echogenicity and thickness) by TVS require, endometrial biopsy remains controversial.

Therefore, if hysteroscopic examination demonstrates the endometrial pattern (echogenicity, vascularity, and thickness) in different PCO cases and correlates it to TVS and histopathology, this would recommend abstinence of endometrial curettage in some PCO patients.

DETAILED DESCRIPTION:
Aim of the work The study aimed to evaluate post menstrual hysteroscopic findings in ovarian PCO and unexplained infertility and correlate them with TVS findings and final histopathologic diagnosis.

Methodology:

1. Study design:

   A cross-sectional study.
2. Setting: Infertility out-patient clinic, Outpatient ultrasonography unit and office hysteroscopy unit of the WWoman'sHealth University Hospital Assiut University.
3. Patients:

   Infertile women in the reproductive age group (18-40 years) whether 1ry or 2ry.
4. Grouping: it will include two groups of infertile women. Group A will consist of 100 PCO infertile women, while group B will consist of 50-unexplained infertility.

Sample size: the previous study could not find endometrial abnormalities hysteroscopy of women with PCOS using of rates. This study will use 100 women aiming to document more accurately the endometrial pattern in women with PCOS.

How is PCO diagnosed in this study? The diagnosis of PCO in this study will use the International evidence-based guideline for the assessment and management of PCOS 2018: The Rotterdam PCOS diagnostic criteria in adults (two of clinical or biochemical hyperandrogenism, ovulatory dysfunction, or polycystic ovaries on ultrasound) and where irregular menstrual cycles and hyperandrogenism are present, highlight that ultrasound is not necessary for diagnosis.

International Evidence-Based Guideline for the Assessment and Management of Polycystic Ovary Syndrome published in 2018 changed the ultrasound criteria from ≥12 to ≥20 antral follicles in an ovary to diagnose PCOS.

PCOS diagnosis is based on oligo-anovulation (OA), biochemical or clinical hyperandrogenism (HA), and polycystic ovary morphology (PCOM) on ultrasound extending across the original 1990 National Institutes of Health (NIH) criteria (OA and HA).

The 2003 Rotterdam criteria (any two of OA, HA, and PCOM) , and the Androgen Excess and Polycystic Ovary Syndrome (AE-PCOS) Society criteria (HA and OA or PCOM or both) .

The Rotterdam criteria are now widely accepted and generate four possible diagnostic PCOS phenotypes in adult women: (A) OA + HA + PCOM, (B) OA + HA, (C) HA + PCOM, and (D) OA + PCOM . The Rotterdam criteria are recommended and endorsed by the 2018 international PCOS evidence-based guideline, which was co-developed based on unprecedented evidence synthesis and best practice methods, by world-leading multidisciplinary clinicians and researchers across 37 societies from 71 countries, with consumer engagement .

Within eight years of menarche, both hyperandrogenism and ovulatory dysfunction are required, with ultrasound not recommended. Ultrasound criteria are tightened with advancing technology. Anti-Müllerian hormone levels are not yet adequate for diagnosis

Data collection:

Demographic data will be collected age, weight, BMI (weight [kg] divided by height in meters squared [m2]), obstetrics and gynecology history (duration of infertility and variability of menstrual cycles), and medications metformin, CC, and tamoxifen. .

TVS findings:

1. International Evidence-Based Guideline for the Assessment and Management of Polycystic Ovary Syndrome published in 2018 Ovarian volume > 10 cm and ≥20antral follicles in an ovary
2. Presence of ovulation or not,
3. endometrial thickness and echognicity,
4. anyadenxal or uterine abnormalities. Doppler U/S. whenever indicated e.g, endometrial mass lesion Hormonal profile assessment: Baseline day 3 serum FSH, LH, Prolactin, TSH. Pre ovulatory urinary LH will be done in all cases.

   Office hysteroscopic examination (2.6 telescopes and 3.2 mm outer sheath): assessment of the following:
   * cervical canal: arborvitae, mucous, any abnormal pathology like a polyp.
   * Endometrium cavity: vascularity, thickness, color, gland openings, any abnormal pathology.
   * Darwish hysterscopic triad: shape, caliber, depth, abnormal pathology, flow patency, bubble flow patency, and peristalsis.

   Endometrial sample by a Novak's curette Histopathologic assessment: will be sent for the routine out-patient Pathology lab to comment on the endometrial pattern and abnormalities.

   Physical and laboratory examinations follicle-stimulating hormone [FSH], LH, thyroid-stimulating hormone [TSH], prolactin, and pre ovulatory LH LH levels of the patients will be measured on day 3 of the menstrual cycle.
5. Ethical considerations:

ELIGIBILITY:
Inclusion Criteria:

1. Reproductive age (18-40).
2. Infertility: 1ry or 2ry.
3. No contraindication for hysteroscopy or histopathology. e.g severe bleeding cervical stenosis.
4. Postmenstrual.

Exclusion Criteria:

* contraindication for hysteroscopy or histopathology. e.g severe bleeding cervical stenosis.
* Non infertility.
* Adolescents and virgins.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
endometrial findings in polycystic and unexplained infertile women | 1 year
  office hysteroscopy to assess endometrial thickness vascularity or any abnormal pathology.

SECONDARY OUTCOMES:
Access to Darwish hysteroscopic triad (DHT) | 1 year
  DHT: a conical area just proximal to the endometrial cavity, its base is the ostium, walls are converging intramural parts of the Fallopian tubes and summit is the narrowist part of the Fallopian tube.

CONTACTS AND LOCATIONS:
Overall Officials: Atef mm Darwish, Study Director — Woman's Health University Hospital
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt